CLINICAL TRIAL: NCT05015608
Title: Clinical Study to Evaluate the Efficacy, Safety and Tolerability of Savolitinib + Osimertinib Versus Pemetrexed + Platinum in Treatment of Patients With NSCLC With MET Amplification
Brief Title: Study on Savolitinib Combined With Osimertinib in Treatment of Advanced NSCLC With MET Amplification
Acronym: SACHI
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-504-00CH3
Record Dates: First submitted 2021-07-30; First posted 2021-08-20 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; osimertinib; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Savolitinib + Osimertinib (Experimental): Savolitinib orally once per day (QD) + Osimertinib orally QD,21day cycles (every 3 weeks)
  Interventions: Drug: Savolitinib + Osimertinib
- Pemetrexed combined with platinum (Active Comparator): Pemetrexed combined with platinumon on Day 1 of 21day cycles (every 3 weeks)
  Interventions: Drug: Pemetrexed + Cisplatin /Carboplatin

INTERVENTIONS:
Drug: Savolitinib + Osimertinib — Subjects will receive Savolitinib orally once per day (QD) + Osimertinib orally QD,21day cycles (every 3 weeks) until disease progression, death, adverse event (AE) leading to discontinuation or withdrawal of consent.
  Arms: Savolitinib + Osimertinib
Drug: Pemetrexed + Cisplatin /Carboplatin — Pemetrexed combined with platinumon on Day 1 of 21day cycles (every 3 weeks)
  Arms: Pemetrexed combined with platinum

SUMMARY:
This study will look at how effective the study drug(Savolitinib combined with Osimertinib) versus Pemetrexed combined with platinum in treatment of patients with locally advanced or metastatic NSCLC with MET amplification after failure of the first-line EGFR inhibitor therapy.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled, open, phase III clinical study to evaluate the clinical efficacy and safety of Savolitinib combined with Osimertinib in treatment of patients with locally advanced or metastatic NSCLC with MET amplification after failure of EGFR inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Fully aware this study and voluntary to sign the informed consent form, and willing and able to comply with the study procedure;
2. Age ≥ 18 and ≤75 years;
3. In accordance with the 8th Edition of TNM staging for lung cancers by International Association for the Study of Lung Cancer and American Joint Committee on Cancer, patients with histologically or cytologically confirmed unresectable and non-suitable for radical concurrent chemoradiotherapy, locally advanced or metastatic (stage IIIB, IIIC or IV) NSCLC;
4. EGFR sensitive mutations prior to the first-line EGFR-TKI therapy;
5. Radiologically documented disease progression after the first-line EGFR-TKI;
6. MET amplification after disease progression following the first-line therapy;
7. Having measurable lesions (in accordance with RECIST 1. 1 criteria);
8. United States Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1;
9. Expected survival >12 weeks;
10. Adequate bone marrow reserve or organ function
11. Female patients of childbearing potential must agree to use effective contraceptive methods from screening period to 4 weeks after discontinuation of the study drug;
12. Male subjects should be willing to agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm. ;
13. Being able to take or swallow the drug orally.

Exclusion Criteria:

1. Patients with positive T790M mutations;
2. Previous treatment for c-MET;
3. Currently having other malignant tumors, or having other infiltrating malignant tumors in the past 5 years.;
4. Previous use of systematic antitumor therapy other than EGFR-TKI for advanced NSCLC;
5. Currently having received antiangiogenic therapy or traditional Chinese medicine with antitumor indication、extensive radiotherapy 、palliative local radiotherapy, a major surgery,or participated in other drug clinical trials and received corresponding tudy drug etc;
6. Currently receiving the potent CYP3A4 inducers or potent CYP1A2 inhibitors within two weeks prior to the start of study treatment;
7. Having not been sufficiently recovered from the toxicity and/or complication resulting from any interventional measure prior to the start of treatment;
8. Clinically significant active infection, including but not limited to tuberculosis, human immunodeficiency virus (HIV) infection (positive HIV1/2 antibody);
9. Active hepatitis B, or active hepatitis C;
10. Acute myocardial infarction, unstable angina pectoris, stroke or transient ischemic attack;
11. Known cancerous thrombus or deep vein thrombosis or uncontrollable hypertension despite the use of drugs;
12. Mean resting corrected QT interval (QTcF) or Any important abnormality in rhythm;
13. Presence of meningeal metastases, spinal cord compression or active brain metastases prior to the start of study treatment;
14. Active gastrointestinal disease or other conditions significantly affecting the absorption, distribution, metabolism or excretion of oral study drug;
15. Lack of compliance with participation in this clinical study or inability to comply with the limitations and requirements of the study, as judged by investigators;
16. Known allergy to the active or inactive ingredient of Savolitinib or Osimertinib;
17. Previous history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis and any active interstitial lung disease;
18. Pregnant or breastfeeding women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 5 months after the last patient enrolled
  Progression-free survival (PFS) using Investigator assessment as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Safety and tolerability | 5 months after the last patient enrolled
  Incidence and nature of treatment emergent adverse events (TEAE), the other safety variables including physical examination, vital signs and laboratory examinations
The objective response rate of the tumor (ORR) | 5 months after the last patient enrolled
  the incidence of confirmed complete response or partial response
The disease control rate (DCR) | 5 months after the last patient enrolled
  the incidence of complete response, partial response and stable disease
Duration of Response (DoR) | 5 months after the last patient enrolled
  the duration between the date the criteria for complete response or partial response was first measured (first record shall prevail) and the date of disease recurrence or progression as objectively recorded
Overall survival (OS) | 5 months after the last patient enrolled
  the time from the date of randomization to the date of death (all causes)
Time to Response (TTR) | 5 months after the last patient enrolled
  the period from the date of randomization to the date when the criteria for complete response or partial response was first measured (first record shall prevail).
PFS | 5 months after the last patient enrolled
  Progression-free survival (PFS) using IRC as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital; Jie Wang, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu S, Wang J, Yang N, Lv D, Chen L, Wu L, Li X, Sun L, Yu Y, Jin B, Yang L, Guo Y, Xu H, Yi T, Zeng A, Dong X, Chen J, Wang Z, Niu H, Cheng Y, Pan P, Deng P, Pan H, Min X, Bai J, Liu L, Zhang T, Li J, Fan S, Shi MM, Mok T, Su W; SACHI Study Group. Savolitinib plus osimertinib versus chemotherapy for advanced, EGFR mutation-positive, MET-amplified non-small-cell lung cancer in China (SACHI): interim analysis of a multicentre, open-label, phase 3 randomised controlled trial. Lancet. 2026 Jan 13:S0140-6736(25)01811-2. doi: 10.1016/S0140-6736(25)01811-2. Online ahead of print. PMID 41544643